CLINICAL TRIAL: NCT06577012
Title: Predicting an Opaque Bubble Layer During Small-Incision Lenticule Extraction Surgery Based on Deep Learning
Brief Title: Potential Risk Factors and Predictive Model Construction of OBL During SMILE
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Yifeng Yu, Deputy chief physician of Ophthalmology center of the Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Other Study IDs: 2024086
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Myopia; Small-incision Lenticule Extraction (SMILE) Surgery
Keywords: small-incision lenticule extraction (SMILE); artificial intelligence; opaque bubble layer
MeSH Terms: conditions — Myopia; Smiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eyes with SMILE surgeries: Eyes with SMILE surgeries which were performed by three surgeons with different experiences.
  Interventions: Procedure: Small incision lenticule extraction

INTERVENTIONS:
Procedure: Small incision lenticule extraction — Small incision lenticule extraction surgeries performed by two Refractive surgery experts (Refractive surgery expert 1: YYF, Associate Professor with 10 years of experience as a refractive surgeon; Refractive surgery expert 2: GF, Associate Professor with 5 years of experience as a refractive surgeon) and a Attending ophthalmologist (XJ, Attending ophthalmologist with 1 year of experience as a refractive surgeon).

SUMMARY:
To explore the prediction of OBL by deep learning model in SMILE surgery

DETAILED DESCRIPTION:
The DL model was used to predict the OBL area during SMILE surgery by identifying the corneal full-view images before laser scanning. The DL model developed may assist surgeons to predict the possible OBL area of patients in advance, so as to adjust some surgical parameters and reduce the formation of OBL, which can avoid negative effects on surgeons' operation and patients' postoperative visual recovery, which has important practical significance.

ELIGIBILITY:
Inclusion Criteria:

* A condition in which the spherical equivalent refractive error of an eye is ≤ -0.50 D when ocular accommodation is relaxed;
* Age ≥18 years;
* Spherical equivalent (SE) ≥ -10.0D;
* Corrected distance visual acuity (CDVA) ≥ 16/20;
* Stable myopia for at least 2 years;
* No contact lenses wearing for at least 2 weeks

Exclusion Criteria:

* The presence or history of eye conditions other than myopia and astigmatism, such as keratoconus or external eye injury;
* A history of eye surgery;
* The presence or history of systemic diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from clinics in ophthalmic center of the second Affiliated Hospital of Nanchang University
Sampling Method: Non-Probability Sample
Enrollment: 4678 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The area of patients with opaque bubble layer in the SMILE surgeries | Day 0
  The area of patients with opaque bubble layer were observed during the SMILE surgeries.

SECONDARY OUTCOMES:
Deep learning model | Day 0
  Predictive performance of deep learning model on the OBL in SMILE surgeries.
ResNet model | Day 0
  Predictive performance of ResNet model on the OBL in SMILE surgeries.
Vgg19 model | Day 0
  Predictive performance of Vgg model on the OBL in SMILE surgeries.
U-net model | Day 0
  Predictive performance of U-net model on the OBL in SMILE surgeries.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No